CLINICAL TRIAL: NCT05243498
Title: Allogenomic Mismatch Score (AMS) Applied to Haplo-identical Donor/Recipient Pairs in Haematopoietic Stem Cell Transplantation
Acronym: AMS-haplo
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Alice AARNINK, PharmD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2021PI066
Record Dates: First submitted 2022-01-13; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Stem Cell Transplantation; Haplo-identical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- no acute GVH, no chronic GVH
  Interventions: Other: Assessment of the Allogenomic Mismatch Score (AMS); Other: Assessment of the optimised Allogenomic Mismatch Score (AMS)
- acute GVH without chronic GVH
  Interventions: Other: Assessment of the Allogenomic Mismatch Score (AMS); Other: Assessment of the optimised Allogenomic Mismatch Score (AMS)
- chronic GVH without acute GVH
  Interventions: Other: Assessment of the Allogenomic Mismatch Score (AMS); Other: Assessment of the optimised Allogenomic Mismatch Score (AMS)
- acute and chronic GVH
  Interventions: Other: Assessment of the Allogenomic Mismatch Score (AMS); Other: Assessment of the optimised Allogenomic Mismatch Score (AMS)

INTERVENTIONS:
Other: Assessment of the Allogenomic Mismatch Score (AMS) — Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient. Roughly, the exome of the donor is aligned to the exome of the recipient, allowing to count the number of variations that will generate a peptide present in the recipient but absent in the donor.
Other: Assessment of the optimised Allogenomic Mismatch Score (AMS) — Optimised Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient, encountering only peptides that can be presented by the donors' MHC (using another layer of algorithm, NetMHCpan).

SUMMARY:
The occurrence of acute and/or chronic GVH (Graf Versus Host disease) for recipients undergoing HSCT (haematopoietic stem cell transplantation) with a geno-identical donor suggests the implication of other systems or genes than those involved in HLA (Human Leukocyte Antigen) compatibility.

In kidney transplantation, it has been shown that the AMS (allogenomic mismatch score) is correlated with the probability of survival of the graft. This AMS reflects the degree of differences between the immunopeptidomes of the recipient and his donor as it is a continuous variable based on the number of nsSNP (non synonymous Single Nucletotide Polymorphism) between the donor and the recipient. Roughly, the exome of the donor is aligned to the exome of the recipient, allowing to count the number of variations that will generate a peptide present in the recipient but absent in in the donor. In this case, peptide presented by the recipient's cells is not part of the donor's immunopeptidome, leading to an activation of the donor's immunocompetent cells toward this antigen, i.e. to alloreactivity that may cause GVL (Graft Versus Leukemia) and/or GVH.

This study aims to highlight significant correlations between the occurrence of acute and/or chronic GVH after haplo-identical stem cell transplantation and the AMS.

This would allow to use the AMS as a predictive factor of acute or chronic GVH, which could be employed to select the best donor for one particular recipient and/or personalize the immunotherapies after transplantation

ELIGIBILITY:
Inclusion Criteria:

* - Recipients who underwent haplo-identical stem cell transplantation in CHRU (Centre Hospitalier Régional et Universitaire) de Nancy
* Recipients transplanted between 03/01/2015 et 01/01/2020
* Recipient older than 18 years old at time of transplant
* Available DNA for the recipient and his donor.

Exclusion Criteria:

* Recipient died within the 6 months following the transplantation without acute GVH (unknown status for one of the measured outcomes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 haplo-identical donor/recipient pairs
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Predictive performance of AMS regarding the occurence of chronic GVH | 12 months after each transplantation
  Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient. Roughly, the exome of the donor is aligned to the exome of the recipient, allowing to count the number of variations that will generate a peptide present in the recipient but absent in the donor. The comparison of AMS will be performed between the groups "presence of cGVH" and "absence of cGVH"

SECONDARY OUTCOMES:
Predictive performance of AMS regarding the occurence of acute GVH | 6 months after each transplantation
  Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient. Roughly, the exome of the donor is aligned to the exome of the recipient, allowing to count the number of variations that will generate a peptide present in the recipient but absent in the donor. The comparison of AMS will be performed between the groups "presence of aGVH" and "absence of aGVH"
Predictive performance of an optimised AMS regarding the occurence of chronic GVH | 12 months after each transplantation
  Optimised Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient, encountering only peptides that can be presented by the donors' MHC (using another layer of algorithm, NetMHCpan). The comparison of optimised AMS will be performed between the groups "presence of cGVH" and "absence of cGVH"
Predictive performance of an optimised AMS regarding the occurence of acute GVH | 6 months after each transplantation
  Optimised Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient, encountering only peptides that can be presented by the donors' MHC (using another layer of algorithm, NetMHCpan). The comparison of optimised AMS will be performed between the groups "presence of aGVH" and "absence of aGVH"
Predictive performance of AMS regarding the occurence of relapse | 12 months after each transplantation
  Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient. Roughly, the exome of the donor is aligned to the exome of the recipient, allowing to count the number of variations that will generate a peptide present in the recipient but absent in the donor. The comparison of AMS will be performed between the groups "relapse" and "no relapse"
Predictive performance of an optimised AMS regarding the occurence of relapse | 12 months after each transplantation
  Optimised Allogenomic Mismatch Score (AMS) is a continuous variable based on the number of nsSNP between the donor and the recipient, encountering only peptides that can be presented by the donors' MHC (using another layer of algorithm, NetMHCpan). The comparison of optimised AMS will be performed between the groups "relapse" and "no relapse"

CONTACTS AND LOCATIONS:
Locations (1):
- Alice Aarnink, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided